CLINICAL TRIAL: NCT06528717
Title: The Role of Maintaining External Carotid Artery Flow in Graft Interposition After Carotid Endarterectomy
Acronym: AGICS
Status: Recruiting | Type: Observational
Sponsor: Institute for Cardiovascular Diseases Dedinje (Other)
Responsible Party: Principal Investigator, Slobodan Pesic, MD, Institute for Cardiovascular Diseases Dedinje
Other Study IDs: 3586
Record Dates: First submitted 2024-07-20; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Carotid Artery Diseases; Stroke; Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ECA flow preserved group: Patients with carotid graft interposition after endarterectomy of the common carotid artery and external carotid artery with preserved flow through the external carotid artery by side-to-end proximal anastomosis.
  Interventions: Procedure: Carotid graft interposition
- Ligated ECA group: Patients with carotid graft interposition and end-to-end anastomoses on the undiseased segments of the common (proximally) and internal (distally) carotid artery, with ligation of the external carotid artery.
  Interventions: Procedure: Carotid graft interposition

INTERVENTIONS:
Procedure: Carotid graft interposition — In patients with extensive atherosclerotic carotid disease, when endarterectomy isn't feasible, replacement of the carotid artery with a graft is needed. Graft interposition can be performed either by end-to-end proximal and distal anastomoses in the undiseased common and internal carotid artery with ligation of the external carotid artery, or by side-to-end proximal anastomosis on the origin of the internal carotid artery and end-to-end distal anastomosis on the internal carotid artery with flow preservation in the external carotid artery.
  Other Names: Carotid artery graft replacement; Carotid replacement with Dacron graft

SUMMARY:
Analyzing results of carotid graft interposition with and without flow preservation through external carotid artery after endarterectomy.

DETAILED DESCRIPTION:
Surgical and endovascular treatment have been shown as effective treatment modalities in symptomatic and asymptomatic patients at high risk of stroke on medical therapy with significant carotid artery stenosis. Eversion carotid endarterectomy (eCEA) has proven effective as a surgical treatment modality. In highly selected instances carotid bypass may be indicated as a bailout procedure or primarily as a preoperatively planned maneuver. Usually, the decision for substitution of carotid bifurcation with a synthetic graft is made due to an extensive, severe atherosclerotic process on the distal part of the extracranial internal carotid artery, the presence of uncontrollable atherosclerotic plaque after endarterectomy, and in cases when an exceptionally thin artery wall remains after endarterectomy.

Several techniques have been described for substituting carotid bifurcation with a synthetic graft. The most common technique involves complete resection and excision of the carotid bifurcation and reconstruction with graft interposition between the undiseased segment of the common carotid artery (CCA) proximally and the internal carotid artery (ICA) distally by creating proximal and distal end-to-end anastomoses. This technique requires ligation and exclusion of the external carotid (ECA) and the superior thyroid artery from circulation. The less common techniques that preserve flow through the external carotid artery are performed as a primary option for treatment without previous endarterectomy and are seldom applied. Currently, there are no recommendations regarding the administration of carotid bypass, nor comparisons of these techniques.

In this study, the investigators are comparing a technique with graft interposition between endarterectomized CCA (creation of side-to-end anastomosis) and the distal segment of the ICA (end-to-end anastomosis) after failure of eCEA to provide technical success with the described common interposition by end-to-end anastomoses proximally and distally. Therefore, the role of flow preservation through the ECA could be defined.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic carotid stenosis (> 50%)
* unilateral asymptomatic carotid stenosis (> 60%)
* bilateral asymptomatic carotid stenosis (> 60%)

Exclusion Criteria:

* carotid restenosis
* "major surgery" in previous 6 months
* previous brain trauma or surgery
* malignant disease
* epilepsy
* carotid artery aneurysm

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent carotid artery surgery due to atherosclerotic symptomatic and asymptomatic disease had graft interposition conducted due to unsuccessful endarterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
periprocedural stroke and death | 30 days
  onset of new neurological deficit or death during perioperative period
myocardial infarction | 30 days
  development of new acute coronary events during perioperative period
stroke ipsilateral to the procedure | through study completion, an average of 2 years
  development of new neurological events that are pathophysiological atributable to the operated side

SECONDARY OUTCOMES:
restenosis rate | through study completion, an average of 2 years
  restenosis after graft placement diagnosed by color Doppler sonographic examination or by multiplanar detection computerized tomography angiography
graft patency | through study completion, an average of 2 years
  primary and primary assisted
patient survival | through study completion, an average of 2 years
  defining cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Srdjan Babic, MD PhD, Study Director — Institute for Cardiovascular Diseases Dedinje
Locations (1):
- Institute for Cardiovascular Diseases Dedinje, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Timaran CH, McKinsey JF, Schneider PA, Littooy F. Reporting standards for carotid interventions from the Society for Vascular Surgery. J Vasc Surg. 2011 Jun;53(6):1679-95. doi: 10.1016/j.jvs.2010.11.122. No abstract available. PMID 21609800